CLINICAL TRIAL: NCT07030517
Title: An Open Label, Multicenter, Phase IV Study of Teclistamab to Evaluate Its Safety in Indian Participants With Relapsed and Refractory Multiple Myeloma Who Have Previously Received at Least 3 Prior Lines of Therapy Including an Immunomodulatory Agent, a Proteasome Inhibitor and an Anti-CD38 Antibody and Have Demonstrated Disease Progression on the Last Therapy
Brief Title: A Study to Assess Safety of Teclistamab in Indian Participants With Relapsed and Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Private Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 64007957MMY4007
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Teclistamab (Experimental): Participants with RRMM eligible for receiving teclistamab will continue to receive study treatment as per the label.
  Interventions: Drug: Teclistamab

INTERVENTIONS:
Drug: Teclistamab — Teclistamab will be administered subcutaneously.
  Other Names: JNJ-64007957

SUMMARY:
The purpose of this study is to assess the safety of teclistamab in routine clinical practice when given as monotherapy in Indian participants with relapsed and refractory multiple myeloma (RRMM) (that is, a blood cancer that comes back after treatment or does not respond to treatment) who have previously received at least 3 prior lines of therapy including an immunomodulatory agent, a proteasome inhibitor and an anti-cluster of differentiation (CD)38 antibody (is a protein that fights infection) and whose disease have progressed on the last therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant with diagnosed RRMM (as per IMWG definitions or investigator's discretion) who have received at least 3 prior lines of therapy including a proteasome inhibitor, an anti-CD 38 antibody and an immunomodulatory agent and have demonstrated disease progression on the last therapy
* Documented evidence of progressive disease on last line of therapy based on investigator's determination of response by IMWG response criteria
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Contraceptive use by female participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. A female participant is eligible to participate if she is not pregnant or breastfeeding, and not a woman of child bearing potential (WOCBP) or is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of less than [<] 1 percent [%] per year), preferably with low user dependency, during the treatment period and for a period of 6 months after the last dose of study treatment and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during study period
* A WOCBP must have a negative highly sensitive serum pregnancy test within 24 hours before the first dose of study treatment

Exclusion Criteria:

* Participants who are not eligible to receive teclistamab as per the locally approved prescribing information
* Received any prior B cell maturation antigen (BCMA)-directed therapy
* Central nervous system (CNS) involvement or clinical signs of meningeal involvement of multiple myeloma. If either is suspected, negative whole brain MRI, and lumbar cytology are required
* Stroke, transient ischemic attack, or seizure within 6 months prior to screening
* Participant had major surgery or had significant traumatic injury within 2 weeks prior to enrollment, or will not have fully recovered from surgery, or has major surgery planned during the time the participant is expected to be treated in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2026-11-03 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAE)s | Up to approximately 2 years 1 month
  An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the intervention under study. TEAEs are AEs with onset during the treatment or that are a consequence of a preexisting condition that has worsened since the first dose of study treatment through the day of last dose plus 30 days or prior to the start of subsequent anticancer therapy, whichever is earlier, or any AE that is considered treatment-related regardless of the start date of the event. TEAEs reported will include all serious and non-serious adverse events.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 2 years 1 month
  ORR is defined as the percentage of participants who have a response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR) or better per investigator assessment according to the International Myeloma Working Group (IMWG) response criteria.
Percentage of Participants With Best Response of Very Good Partial Response (VGPR) or Better | Up to approximately 2 years 1 month
  VGPR or better response rate is defined as the percentage of participants who achieve a response of VGPR or better response (sCR, CR and VGPR) as per investigator assessment according to the IMWG response criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Private Limited Clinical Trial, Study Director — Johnson & Johnson Private Limited
Locations (11):
- India (11):
  - M S Ramaiah Medical College and Hospital, Bangalore
  - St. Johns Medical College And Hospital, Bengaluru
  - Post Graduate Institute of Medical Education And Research PGIMER, Chandigarh
  - Bhagwan Mahaveer Cancer Hospital & Research Centre, Jaipur
  - Tata Medical Center, Kolkata
  - Tata Memorial Hospital, Mumbai
  - KIMS-Kingsway Hospitals, Nagpur
  - All India Institute of Medical Sciences, New Delhi
  - Rajiv Gandhi Cancer Institute & Research Centre, New Delhi
  - Christian Medical College, Ratnagiri Kilminnal
  - Regional Cancer Centre, Thiruvananthapuram

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency